CLINICAL TRIAL: NCT02650973
Title: A Randomized, Single-Blind, Crossover Study to Assess the Pharmacokinetic and Pharmacodynamic Bioequivalence of CHS-1701 (Coherus Pegfilgrastim) With Neulasta® in Healthy Subjects
Brief Title: Study to Assess the Pharmacokinetic and Pharmacodynamic Bioequivalence of CHS-1701 With Neulasta
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Coherus Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: CHS-1701-05
Record Dates: First submitted 2016-01-05; First posted 2016-01-08 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Healthy
Keywords: Bioequivalence
MeSH Terms: interventions — pegfilgrastim

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sequence A (Experimental): 3 doses of CHS-1701 or Neulasta, random order
  Interventions: Drug: CHS-1701; Drug: Pegfilgrastim
- Sequence B (Experimental): 3 doses of CHS-1701 or Neulasta, random order
  Interventions: Drug: CHS-1701; Drug: Pegfilgrastim
- Sequence C (Experimental): 3 doses of CHS-1701 or Neulasta, random order
  Interventions: Drug: CHS-1701; Drug: Pegfilgrastim

INTERVENTIONS:
Drug: CHS-1701
Drug: Pegfilgrastim
  Other Names: Neulasta

SUMMARY:
This is a randomized, single-blind, 3-period crossover study in healthy subjects to assess PK, PD, and safety (including immunogenicity) of a single 6mg subcutaneous injection of CHS-1701 (Coherus pegfligrastim) or 6mg SC dose of Neulasta (pegfilgrastim) given during each period.

DETAILED DESCRIPTION:
This is a randomized, single-blind, 3-period crossover study in healthy subjects to assess PK, PD, and safety (including immunogenicity) of a single 6mg subcutaneous injection of CHS-1701 or 6mg SC dose of Neulasta given during each period.

The screening period may occur up to 28 days prior to the confinement period. After screening, eligible subjects will be randomly assigned to one of three possible treatment sequences. Treatments will be spaced by not less than 28 days.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female of ages 18 to 45 inclusive
2. Body weight > 50 kg (110 lb.) and body mass index between 18 and 28 kg/m2 inclusive
3. Medically healthy with clinically insignificant findings based on medical history, 12-lead ECG, and physical examination
4. Negative urine pregnancy test in women of childbearing potential

Exclusion Criteria:

1. Previous exposure to pegfilgrastim or filgrastim
2. Current or previous cancer, diabetes, or any clinically significant cardiovascular, metabolic, endocrine, renal, hepatic, gastrointestinal, hematologic, respiratory, dermatological, neurological, gynecologic, psychiatric, or other disorder
3. History of chronic or acute respiratory illness within the past 3 months
4. Positive urine drug or alcohol screen or unwillingness to abstain from alcohol or recreational drugs for the duration of study participation
5. No prescription or nonprescription drugs during the study
6. Participation in an investigational clinical study within 30 days prior to screening
7. History of known clinically significant drug and/or food allergies, including allergic reaction to latex

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 122 (Actual)
Dates: Start 2016-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Bioequivalence as measured by PK and PD | 84 Days
  The primary objective of this study is to assess the bioequivalence of CHS-1701 with Neulasta® based on the pharmacokinetics (PK) of pegfilgrastim and the pharmacodynamic (PD) response as measured by absolute neutrophil count (ANC)

SECONDARY OUTCOMES:
PK Profile: Cmax | 84 Days
  Characterization of the PK profile of CHS-1701 using standard parameters of maximum plasma concentration (Cmax)
PK Profile: tmax | 84 Days
  Characterization of the PK profile of CHS-1701 using standard parameters of time to maximum plasma concentration (tmax)
PK Profile: AUC0-t | 84 Days
  Characterization of the PK profile of CHS-1701 using standard parameters of area under the plasma concentration versus time curve calculated from 0 to the last measurable observation (AUC0-t)
PK Profile: t1/2 | 84 Days
  Characterization of the PK profile of CHS-1701 using standard parameters of terminal elimination half-life (t1/2)
Safety Profile as assessed by clinical adverse events (AEs), laboratory variables, vital signs, incidence of antidrug antibodies (ADAs), and local injection site reactions (ISRs) | 84 Days
  Characterization of the safety profile and tolerance of CHS-1701, as assessed by clinical adverse events (AEs), laboratory variables, vital signs, incidence of antidrug antibodies (ADAs), and local injection site reactions (ISRs).

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Finck, MD, Study Director — Coherus BioSciences
Locations (4):
- United States (4):
  - WCCT, Cypress, California
  - Medpace CPU, Cincinnati, Ohio
  - ICON, San Antonio, Texas
  - Spaulding, West Bend, Wisconsin

REFERENCES:
- [Derived] Civoli F, Finck B, Tang H, Hodge J, O'Kelly H, Vexler V. Biosimilar Pegfilgrastim-cbqv Demonstrated Similar Immunogenicity to Pegfilgrastim in Healthy Subjects Across Three Randomized Clinical Studies. Adv Ther. 2022 Mar;39(3):1230-1246. doi: 10.1007/s12325-021-02024-x. Epub 2022 Jan 16. PMID 35034311
- [Derived] Finck B, Tang H, Civoli F, Hodge J, O'Kelly H, Vexler V. Pharmacokinetic and Pharmacodynamic Equivalence of Pegfilgrastim-cbqv and Pegfilgrastim in Healthy Subjects. Adv Ther. 2020 Oct;37(10):4291-4307. doi: 10.1007/s12325-020-01459-y. Epub 2020 Aug 13. PMID 32789809